CLINICAL TRIAL: NCT00005370
Title: Longitudinal Study of Cortisol and Pulmonary Function
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4261; R01HL049869 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-11

CONDITIONS: Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To conduct a longitudinal study of the relationship between the rate of decline of pulmonary function and measurements of cortisol concentration and excretion in a sample of middle-aged and older men and their wives. The study tested the hypothesis that persons whose plasma cortisol concentrations were relatively low, albeit within the normal range, were predisposed to excessively rapid deterioration of pulmonary function during aging.

DETAILED DESCRIPTION:
BACKGROUND:

It was hoped that the study would provide important insights into the pathogenesis of chronic obstructive pulmonary disease with potential implications for prevention and early therapeutic intervention.

DESIGN NARRATIVE:

All subjects participating in the Normative Aging Study were recruited for the study at the time of their next scheduled examination. Twenty-four hour urinary excretion of free cortisol, morning serum cortisol concentration, and pre- and post-bronchodilator spirometric indices were measured. For the 700 subjects who were recruited during years one and two of the study, these measurements were repeated when subjects returned for their next triennial examination in years four and five of the study. Respiratory illness and smoking questionnaire data, total and differential leukocyte counts, and methacholine inhalation challenge test data were also available at both time points. The specific aims of the study were to examine: (1) the cross-sectional relationship between level of pulmonary function and both morning serum cortisol concentration and 24-hour urinary free cortisol excretion; (2) the relationship between the rate of decline of pulmonary function during the follow-up interval and these measurements of cortisol concentration and excretion; (3) whether these relationships were modified by smoking history, blood total leukocyte count, methacholine airway responsiveness, or other characteristics; and (4) the stability over time of serum cortisol concentration and urinary cortisol excretion in this aging population.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-04; Study Completion 1999-03 (Actual)